CLINICAL TRIAL: NCT02708849
Title: The Sustained Effects of Ketamine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1501015203
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Ketamine; Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine plus lamotrigine (Experimental)
  Interventions: Drug: Ketamine; Drug: Lamotrigine
- ketamine plus placebo (Placebo Comparator)
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — The subanesthetic dose of ketamine (0.23mg/kg bolus followed by 0.58mg/kg infusion over approximately 60 minutes) will be administered via intravenous infusion
Drug: Lamotrigine — lamotrigine (300 mg oral dose) or the matched-placebo control about 2-hours prior to the start of the infusion of ketamine
  Arms: Ketamine plus lamotrigine
Drug: Placebo — oral dose placebo
  Arms: ketamine plus placebo

SUMMARY:
The purpose of the study is to characterize the effects of a single, sub-anesthetic dose of ketamine in rs-fMRI in healthy subjects. Post-ketamine rs-fMRI data will demonstrate a pattern of increased global brain connectivity (GBC) in fronto-temporal cortex.

DETAILED DESCRIPTION:
In this study, healthy participants will be randomized into one of two parallel groups: (a) open-label ketamine and active lamotrigine, or (b) open-label ketamine with a matched-placebo control (i.e., sugar pill). All participants will complete a baseline rs-fMRI approximately 1-week prior to the ketamine infusion and a follow-up rs-fMRI 24-hours post-infusion. The subanesthetic dose of ketamine (0.23mg/kg bolus followed by 0.58mg/kg infusion over approximately 60 minutes) will be administered via intravenous infusion to occur during the MRS scan. Participants will be administered lamotrigine (300 mg oral dose) or the matched-placebo control about 2-hours prior to the start of the infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 21-65 years. Females will be included if they are not pregnant and agreed to utilize a barrier method contraceptive (e.g., condom or diaphragm with spermicide) tubal ligation, abstinence, or partner with vasectomy) or if post-menopausal for at least 1 year, or surgically sterile.
* Able to provide written informed consent according to Yale HIC guidelines.
* Agree to refrain from elective surgeries (including dental) for a 2-week period following study drug.
* Able to read and write English as a primary language.

Exclusion Criteria:

* Personal history of mood, anxiety, or psychotic axis I DSM-IV disorders confirmed after comprehensive psychiatric evaluation.
* Any history of serious medical or neurological illness.
* Any signs of major medical or neurological illness on examination or as a result of ECG screening or laboratory studies.
* A first-degree family member with history of schizophrenia.
* Lifetime history of psychoactive substance or alcohol dependence or substance or alcohol abuse (other than nicotine or caffeine abuse), or drinking more that 5 drinks/week during the last year.
* Abnormality on physical examination. A subject with a clinical abnormality may be included only if the study physician considers the abnormality will not introduce additional risk factors and will not interfere with the study procedure (e.g. uncontrolled hypertension, hyperthyroidism, or hypothyroidism will be excluded).
* A positive pre-study (screening) urine drug screen or, at the study physician's discretion on any drug screens given before the scans.
* Pregnant or lactating women or a positive urine pregnancy test for women of child-bearing potential at screening or prior to any imaging day.
* Positive HIV or Hepatitis B/C tests. This test will take place at the screening visit. Subjects will be invited back either for their next study visit or for a HIV/Hep debriefing session. A study clinician will inform them in person of the results. They will be given access to counselling and advised of the appropriate next steps.
* Has received either prescribed or over-the-counter (OTC) centrally active medicine or herbal supplements within the week prior to the MRI scan. Subjects who have taken OTC medication or herbal supplements may still be entered into the study, if, in the opinion of the principal/co-investigator, the medication received will not interfere with the study procedures or compromise safety.
* Any history indicating learning disability, mental retardation, or attention deficit disorder.
* Known sensitivity to ketamine.
* Known sensitivity to lamotrigine.
* Body weight of 250 pounds or greater.
* History of claustrophobia.
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI screening questionnaire.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Resting blood pressure lower than 90/60 or higher than 150/90, or resting heart rate lower than 45/min or higher than 100/min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-06; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Abdallah, MD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Plus Lamotrigine | Ketamine Plus Placebo
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Plus Lamotrigine | Ketamine Plus Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Due to the small sample size in each arm, we did not analyze the ages separately and baseline measures were not provided to protect confidentiality of participants. We provided date for the analysis of age for the total number of participants.
  years | NA (NA) — data was not analyzed due to the small sample size | NA (NA) — data was not analyzed due to the small sample size | 40 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Post-Ketamine Rs-fMRI Data
Description: 24 hours post infusion fMRI data
Time Frame: 24 hours
Population: Imaging data were not extracted to protect confidentiality of participants.
Arm/Group | Ketamine Plus Lamotrigine | Ketamine Plus Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Global Brain Connectivity
Description: Participants will be randomized into one of two parallel groups-ketamine+lamotrigine or ketamine+placebo-and will complete pre- and post-ketamine rs-fMRI.
  The hypothesis is that post-ketamine rs-fMRI data will demonstrate a pattern of increased global brain connectivity (GBC) in fronto-temporal cortex.
  Insufficient number of participants for data collection.
Time Frame: 24 hours
Population: Insufficient number of participants for data collection
Arm/Group | Ketamine Plus Lamotrigine | Ketamine Plus Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Ketamine Plus Lamotrigine | Ketamine Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT02708849/Prot_SAP_000.pdf